CLINICAL TRIAL: NCT06614140
Title: A Phase I/IIb Study of Personalized Neoantigen Peptide-Based Cancer Vaccine for Patients with Solid Tumors
Brief Title: Personalized Neoantigen Cancer Vaccine for Patients with Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Seqker Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SQK01-001
Record Dates: First submitted 2024-09-19; First posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Cancer; Solid Tumor, Adult
Keywords: neoantigen; vaccine; personalized; cancer; peptide
MeSH Terms: conditions — Neoplasms | interventions — poly ICLC

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Personalized Neoantigen Peptide Vaccine with Poly-ICLC and Checkpoint Inhibitors (Experimental): Participants will receive a personalized neoantigen peptide vaccine based on tumor-specific mutations identified through genomic analysis. The treatment has three phases:
  Preparation Phase: Poly-ICLC, an immune adjuvant, is given intramuscularly twice weekly for four weeks before the first vaccine dose to enhance immune readiness.
  Treatment Phase: The neoantigen vaccine is administered with Poly-ICLC on days 1, 4, 8, 15, and 22. A checkpoint inhibitor (e.g., anti-PD-1 or anti-PD-L1) will be introduced after neoantigen-specific T cell responses are detected to counteract immune exhaustion. Booster injections are given at weeks 12 and 20.
  Follow-up Phase: Checkpoint inhibitors (per standard regimen) and Poly-ICLC (twice monthly) will be continued to maintain the immune response. Safety, immune activity, and clinical outcomes will be closely monitored.
  Interventions: Biological: Personalized Neoantigen Peptide Vaccine with Poly-ICLC and Checkpoint Inhibitors

INTERVENTIONS:
Biological: Personalized Neoantigen Peptide Vaccine with Poly-ICLC and Checkpoint Inhibitors — This intervention involves a personalized neoantigen peptide vaccine composed of peptides containing tumor-specific mutations, such as SNVs, indels, and frameshift mutations. Neoantigens are selected based on criteria that enhance expression and immunogenicity.
  The vaccine is administered alongside Poly-ICLC, a TLR3 agonist, to enhance immune activation. After the initial vaccine doses, checkpoint inhibitors (e.g., anti-PD-1 or anti-PD-L1) are introduced once neoantigen-specific T-cell responses are detected, preventing immune exhaustion and sustaining a strong immune response.
  During the follow-up phase, both checkpoint inhibitors and Poly-ICLC are continued to maintain immune activity and ensure a lasting anti-tumor effect.

SUMMARY:
This clinical trial aims to evaluate the safety, immunogenicity, and preliminary efficacy of a personalized neoantigen peptide vaccine in patients with advanced cancer or at high risk of recurrence. The study is designed for patients whose tumors have specific mutations identifiable through genomic sequencing. These mutations, known as neoantigens, are unique to each patient's cancer and serve as the target for the personalized vaccine.

Eligible patients will undergo genomic analysis, including whole exome sequencing and RNA sequencing, to identify these neoantigens. A custom peptide vaccine will then be produced and formulated to target these neoantigens. The trial consists of a preparation phase, a treatment phase with priming and booster vaccinations, and a follow-up/maintenance period of one year. The study will assess immune responses, clinical efficacy, and potential toxicities. By leveraging the immune system's ability to recognize and attack cancer cells, this vaccine aims to provide a new treatment option for patients with limited alternatives.

DETAILED DESCRIPTION:
This Phase Ib/II, open-label, single-center study investigates the safety, immunogenicity, and preliminary efficacy of a personalized neoantigen peptide vaccine in patients with advanced cancer or high risk of recurrence. The trial aims to enroll 15-35 eligible patients and is divided into three phases: preparation, treatment, and follow-up.

Preparation Phase: Patients undergo genomic analysis using whole exome sequencing and RNA sequencing to identify specific neoantigens from their tumor tissues. Based on these findings, a personalized neoantigen peptide vaccine is produced and formulated. Poly-ICLC, an immune adjuvant, is administered intramuscularly twice weekly for four weeks prior to the first vaccine dose to enhance immune readiness.

Treatment Phase: The neoantigen peptide vaccine is administered alongside Poly-ICLC on days 1, 4, 8, 15, and 22. A checkpoint inhibitor (e.g., anti-PD-1 or anti-PD-L1) will be introduced once neoantigen-specific T cell responses are detected, to prevent immune exhaustion and sustain the immune response. Booster injections of the neoantigen vaccine are scheduled for weeks 12 and 20. Immune responses and adverse events will be closely monitored throughout this phase.

Follow-up Phase: During the follow-up phase, checkpoint inhibitors (administered per standard regimen) and Poly-ICLC (administered twice monthly) will be continued to maintain immune activity and ensure a lasting anti-tumor response. Safety, immune activity, and clinical outcomes will be closely monitored over a one-year period.

The primary endpoints include safety and immunogenicity, measured by adverse event monitoring and T-cell activation assays. Secondary endpoints will assess clinical efficacy, including tumor response rates, progression-free survival, and overall survival. Exploratory endpoints will involve biomarker analysis and immune profiling to correlate clinical outcomes with specific immune responses.

This study aims to validate the hypothesis that personalized neoantigen peptide vaccines, in combination with immune adjuvants and checkpoint inhibitors, can elicit strong immune responses and improve clinical outcomes in patients with advanced or high-risk recurrent cancers, especially where standard therapies have failed.

ELIGIBILITY:
Inclusion Criteria:

Cancer patients will be selected from those receiving treatment at the Cancer Center, Vejthani Hospital. All participants must meet the following criteria:

1. Cancer patients must be aged 18 years or older.
2. Patients must provide informed consent and voluntarily agree to participate in the study.
3. Patients must have an estimated life expectancy of at least 6 months.
4. Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-1 and normal functioning of internal organs.
5. Patients must have been diagnosed with cancer based on clinical presentation and confirmed by pathological evidence, including diagnostic imaging.
6. Specific criteria for the cancer type under study:

   * Advanced-stage cancer: No available standard treatment, resistant to standard therapies, and/or the patient is ineligible or refuses standard treatments.
   * Early-stage cancer with high recurrence risk: Even after surgery and/or radiation therapy and completion of standard treatment, the cancer has a high risk of recurrence, and there is no clear adjuvant treatment available.
7. Patients must have tumor tissue suitable for analysis and production of neoantigen peptides.
8. For advanced-stage cancer (not in the adjuvant setting), patients must have radiologic evidence that can be used to assess response according to mRECIST1.1 criteria for solid tumors.
9. Patients must have normal liver, kidney, and laboratory function, as indicated by the following criteria:

   * Lymphocyte count ≥ 800 cells/µL
   * Neutrophil count ≥ 1,500 cells/µL
   * Platelet count ≥ 150,000 cells/µL
   * AST ≤ 2.5 times the upper limit of normal (ULN)
   * ALT ≤ 2.5 times the ULN
   * Total bilirubin ≤ 1.5 times the ULN
   * Serum creatinine ≤ 1.5 times the ULN
10. Patients must agree to avoid pregnancy or causing pregnancy, according to the following:

    * Female patients not of childbearing potential, defined as those who have had a hysterectomy and/or bilateral oophorectomy, have experienced menopause for more than 12 months, or are aged over 60.
    * Female patients of childbearing potential must have a negative pregnancy test during the preparation phase and before receiving the first dose of the vaccine. They must also agree to use effective contraception from the preparation phase until 120 days after the last treatment.
    * Male patients must agree to use effective contraception from the preparation phase until 180 days after the last treatment.

Exclusion Criteria:

Cancer patients will not be eligible to participate in the study if they meet any of the following conditions:

1. Patients with a known history of allergy to peptide vaccines.
2. Patients with a history of autoimmune disease.
3. Patients who have received chemotherapy or radiation therapy less than 4 weeks prior to enrollment or as determined by the physician. This also includes patients with unresolved side effects from previous treatment graded ≥2 (CTCAE v4.0).
4. Patients with cancer that has metastasized to the brain or central nervous system, unless they have been treated and the metastases are controlled, and have been off steroids for at least 4 weeks.
5. Patients with a history of another malignancy within the past 2 years, except for locally treated basal cell or squamous cell skin cancer.
6. Patients with a history of Human Immunodeficiency Virus (HIV) infection.
7. Patients with a history of Hepatitis B or C infection. For those without prior history, screening will be conducted. Patients who test positive for Hepatitis B (HBsAg) or Hepatitis C (HCV) will be excluded unless:

   * Hepatitis B is controlled with antiviral treatment, as evidenced by an undetectable viral load.
   * Hepatitis C has been treated and the viral load is undetectable.
8. Patients with symptomatic or uncontrolled heart disease, including unstable angina, acute myocardial infarction, heart failure (New York Heart Association Class III or IV), or arrhythmias requiring treatment.

   * Patients with pacemakers may be eligible if their heart rhythm has been stable for at least one month before receiving the neoantigen peptide vaccine.
9. Patients who have received live attenuated or killed vaccines within 28 days prior to the first dose of the neoantigen peptide vaccine.
10. Patients receiving immunosuppressive drugs or corticosteroids at a dose of more than 10 mg of prednisolone (except for inhaled or intranasal corticosteroids) within the last 4 weeks before enrollment.
11. Patients with underlying medical conditions that may interfere with the efficacy or safety of the peptide vaccine.
12. Pregnant or breastfeeding patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2022-11-24 (Actual); Primary Completion 2025-08-15 (Estimated); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
Safety of the Personalized Neoantigen Peptide Vaccine | From the start of treatment through the follow-up phase (up to 18 months).
  Safety will be assessed by monitoring the incidence, frequency, severity, and type of adverse events (AEs) and serious adverse events (SAEs) throughout the study, graded according to the Common Terminology Criteria for Adverse Events (CTCAE).
Immunogenicity of the Personalized Neoantigen Peptide Vaccine | From the start of treatment through the follow-up phase (up to 18 months).
  Immunogenicity will be measured by evaluating T-cell responses specific to the neoantigen peptides in the peripheral blood of patients. Assays such as ELISpot and flow cytometry will be used to quantify neoantigen-specific T cells before and after vaccine administration to assess the vaccine's ability to stimulate an immune response.

SECONDARY OUTCOMES:
Tumor Response Rate (Objective Response Rate) based on mRECIST 1.1 | From the start of treatment until disease progression or up to 18 months, whichever occurs first.
  Tumor response rate will be assessed using mRECIST 1.1 criteria, which includes the objective measurement of tumor shrinkage or growth.
Progression-Free Survival (PFS) | From the start of treatment until disease progression, death, or up to 24 months, with follow-up beyond the primary study time frame for long-term evaluation.
  PFS will be measured as the time from the start of treatment to the first documented disease progression, or death, whichever occurs first.
Overall Survival (OS) | From the start of treatment until death, last follow-up, or up to 5 years, with long-term follow-up beyond the primary study time frame to assess overall survival trends.
  OS will measure the length of time from the start of treatment until death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Vejthani Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No